CLINICAL TRIAL: NCT01154296
Title: Project Aware: HIV Rapid Testing & Counseling in STD Clinics in the U.S. -- an Adaptation of CTN 0032
Brief Title: HIV Rapid Testing & Counseling in Sexually Transmitted Disease (STD) Clinics in the U.S.
Acronym: Aware
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); University of Pittsburgh (Other); University of California, San Francisco (Other); Oregon Health and Science University (Other); Medical University of South Carolina (Other); Research Foundation for Mental Hygiene, Inc. (Other); Duke University (Other); The Emmes Company, LLC (Industry); San Francisco Department of Public Health (Other Government); University of California (Other); Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Lisa Metsch, Stephen Smith Professor of Sociomedical Sciences and Chair, Department of Sociomedical Sciences, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: AAAK3153; 1RC2DA028973-01 (NIH)
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Results first posted 2014-09-29 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: HIV/AIDS; Sexually Transmitted Infections
Keywords: HIV; Rapid Testing; Counseling; STD; U.S.
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rapid HIV Testing w/ Counseling (Group 1) (Experimental): Individuals who screen as eligible will complete written informed consent procedures, be enrolled, be tested for STIs, and be asked to complete a baseline assessment using audio computer-assisted self interview (ACASI). Then participants randomized to group 1 will receive rapid HIV testing and RESPECT-2 counseling.
  Interventions: Behavioral: RESPECT-2 Counseling
- Rapid HIV Testing & Information Only (Group 2) (No Intervention): Individuals who screen as eligible will complete written informed consent procedures, be enrolled, be tested for STIs, and be asked to complete a baseline assessment using audio computer-assisted self interview (ACASI). Then participants randomized to group 2 will receive rapid HIV testing with information only.

INTERVENTIONS:
Behavioral: RESPECT-2 Counseling — Specifically designed for use with the rapid HIV test, involves a brief (approximately 20-40 minute) counseling session which includes an orientation to the rapid testing procedure, an explanation of the testing window period, routes of HIV transmission and the meaning of test results, a personalized exploration of risk, the creation of a risk-reduction plan, identification of sources for support and referrals, and HIV test results.
  Other Names: RESPECT-2 Protocol
  Arms: Rapid HIV Testing w/ Counseling (Group 1)

SUMMARY:
Project Aware is a randomized controlled clinical trial in which individuals seeking medical or health services at sexually transmitted disease (STD) clinics are recruited to participate in a multi-center HIV testing and counseling study. The investigators will assess the relative effectiveness and cost-effectiveness of (1) on-site HIV rapid testing with brief, participant-tailored prevention counseling vs. (2) on-site HIV rapid testing with information only. The investigators will evaluate the effect of counseling on one primary outcome: STI incidence. Secondary outcomes will be reduction of sexual risk behaviors, substance use during sex (i.e., being under the influence during sex) and cost and cost effectiveness of counseling and testing. Participants will be assessed for sexually transmitted infections, HIV testing history and sexual and drug use risk behaviors at baseline and at 6-months follow-up. Approximately 5,000 individuals seeking medical or health services from approximately 9 STD clinics throughout the United States will be randomized. These individuals will be 18 years of age or older and efforts will be made to recruit a sample of study participants that reflects the proportion of minorities and gender in the STD clinic performance sites from which the investigators are recruiting.

DETAILED DESCRIPTION:
An estimated 56,300 Americans are newly infected with HIV every year. In addition, of the more than one million Americans living with HIV, approximately one-fifth do not know they are infected. Identifying these individuals is among the biggest challenges for HIV prevention in the United States. Early diagnosis of such individuals, combined with prevention counseling and provision of health care, could decrease the spread of HIV and improve the survival of HIV-infected persons.

The recent introduction of rapid HIV testing offers a critical public health screening approach for facilitating earlier diagnoses of HIV infection. Rapid tests permit a sensitive and specific, fast, simple, minimally invasive, and cost-effective method to screen for HIV.

Project Aware expands on the CDC's Project RESPECT-2 study that was an expansion of the RESPECT study (a randomized controlled trial conducted in STD clinics in the mid-1990s before the advent of highly active antiretroviral therapy and before the advent of rapid testing). Project RESPECT demonstrated that a 2-session, client centered counseling session based on behavioral theory with HIV testing was superior to a program with HIV testing and information only. This project showed that the counseling arm had significant reduction of STIs compared to those in the information arm. However, RESPECT did not include men who have sex with men (who account for 53% of all new HIV infections in the U.S.) and did not examine the cost effectiveness of the intervention. RESPECT-2 did include MSM, but it only compared a 1-session counseling session with rapid testing to 2-session counseling with traditional testing and did not address the question of whether counseling and testing is more effective than testing alone.

Project Aware combines the RESPECT-2 counseling approach by adapting the HIV Rapid Testing and Counseling in Drug Abuse Treatment Study (CTN 0032), a NIDA-sponsored randomized controlled clinical trial being conducted in the NIDA Clinical Trials Network (CTN) to sexually transmitted disease (STD) clinics to provide important and timely data on the effect of counseling in high-risk populations tested in health care settings. In this adaptation of CTN 0032, we will assess the relative effectiveness of (1) on-site HIV rapid testing with brief, participant-tailored prevention counseling vs. (2) on-site HIV rapid testing with information only (as recommended in the CDC guidelines). Secondary outcomes are reduction of sexual risk behaviors, substance use during sex (i.e., being under the influence during sex) and cost and cost effectiveness of counseling and testing. Participants (approximately 5,000 from 9 STD clinics) will be assessed for STIs, HIV testing history and sexual and drug use risk behaviors at baseline and at 6-months follow-up. The battery of STI tests will screen for Neisseria gonorrhea (GC), Chlamydia trachomatis (CT), Trichomonas vaginalis, Herpes Simplex 2 (HSV-2) and Treponema pallidum (syphilis). HIV test results that yield a reactive result will receive a confirmatory HIV blood test that day, with results delivered 5-10 days later. All participants will be randomized into one of two arms: Group 1- HIV testing and brief, client-centered counseling or Group 2- HIV testing and information only. Group 1 will receive a rapid HIV test with brief prevention counseling that addresses risk reduction based on an evidence-based counseling approach (RESPECT-2 counseling), while Group 2 will receive a rapid HIV test with information only.

The primary outcome will be analyzed using logistic regression for the binary outcome, new diagnoses of STIs (Yes/No). The logistic regression analysis will predict 6-month STI incidence as a function of randomization group controlling for the baseline incidence of STI. ANCOVA will be used for the secondary continuous outcomes, number of sexual risk behaviors and number of sexual episodes involving substance use. Costs will be compared based on study records supplemented by site-level data collection. Primary analyses will be performed under intent-to-treat (ITT) criteria.

ELIGIBILITY:
Inclusion Criteria:

* Site Eligibility:

  1. high rates of STIs and HIV in their geographic target area,
  2. sufficient number of patients so that they would be able to recruit the required 556 participants over the study time period,
  3. prior participation in research and clinical studies, and
  4. previous collaboration with investigators.
* Participant eligibility:

  1. be seeking medical or health services at the participating STD clinic,
  2. be at least 18 years old,
  3. report being HIV-negative or status unknown,
  4. provide informed consent,
  5. provide locator information,
  6. be able to communicate in English,
  7. agree to be tested for STIs/STDs and HIV;
  8. sign a HIPAA form and/or medical record release form to permit medical record abstraction of HIV and STI/STD tests, results and treatment; and
  9. report living in the vicinity of the clinic and being able to return to the clinic for the 6-month follow-up visit.

Exclusion Criteria:

* Sites:

  1. low rates of STIs and HIV in their geographic target area,
  2. insufficient number of patients to meet study needs of 556 per site
  3. no prior participation in research and clinical studies, and
  4. no previous collaboration with investigators.
* Participants:

  1. Not seeking medical or health services at the participating STD clinic,
  2. under 18 years old,
  3. HIV positive,
  4. unwilling to provide Informed Consent,
  5. refuse to provide locator information,
  6. not able to communicate in English,
  7. Disagree to be tested for STIs/STDs and/or HIV, and
  8. unwilling to sign a HIPAA form and/or medical record release form to permit medical record abstraction of HIV and STI/STD tests, results and treatment,
  9. report living out of the vicinity and unable to return to the clinic for the 6-month follow-up visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5012 (Actual)
Dates: Start 2010-04; Primary Completion 2011-07 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa R. Metsch, Ph.D., Principal Investigator — University of Miami; Grant N Colfax, M.D., Principal Investigator — San Francisco Department of Public Health
Locations (9):
- United States (9):
  - Los Angeles Gay & Lesbian Center, Los Angeles, California
  - San Francisco Department of Public Health, San Francisco, California
  - Whitman-Walker Clinic, Washington D.C., District of Columbia
  - Duval County Health Department, Jacksonville, Florida
  - Miami-Dade County Health Department, Miami, Florida
  - Multnomah County Health Department, Portland, Oregon
  - Allegheny County Health Department, Pittsburgh, Pennsylvania
  - Richland County Health Department, Colombia, South Carolina
  - Public Health Seattle & King County, Seattle, Washington

REFERENCES:
- [Result] Metsch LR, Feaster DJ, Gooden L, Schackman BR, Matheson T, Das M, Golden MR, Huffaker S, Haynes LF, Tross S, Malotte CK, Douaihy A, Korthuis PT, Duffus WA, Henn S, Bolan R, Philip SS, Castro JG, Castellon PC, McLaughlin G, Mandler RN, Branson B, Colfax GN. Effect of risk-reduction counseling with rapid HIV testing on risk of acquiring sexually transmitted infections: the AWARE randomized clinical trial. JAMA. 2013 Oct 23;310(16):1701-10. doi: 10.1001/jama.2013.280034. PMID 24150466
- [Derived] Alcaide ML, Feaster DJ, Duan R, Cohen S, Diaz C, Castro JG, Golden MR, Henn S, Colfax GN, Metsch LR. The incidence of Trichomonas vaginalis infection in women attending nine sexually transmitted diseases clinics in the USA. Sex Transm Infect. 2016 Feb;92(1):58-62. doi: 10.1136/sextrans-2015-052010. Epub 2015 Jun 12. PMID 26071390

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individuals seeking services at 9 sexually transmitted disease (STD) clinics across the U.S. were recruited, screened and randomized between April 2010 - December 2010.
Pre-assignment Details: Study personnel made 14,948 approaches to STD clinic patients; some were approached multiple times. Of the 6,239 consenting to be screened, 5028 were eligible (80.6%); 16 of these were not randomized due to: decision to decline (n=3), not returning (n=11), not testing with HIV/STD battery (n=1) and not completing baseline activities (n=1).
Period: Randomization and Intervention
Arm/Group | Rapid HIV Testing w/ Counseling (Group 1) | Rapid HIV Testing & Information Only (Group 2)
Started | 2505 | 2507
Completed | 2500 | 2505
Not Completed | 5 | 2
Not completed — Decided to decline | 1 | 1
Not completed — Declined by staff | 1 | 0
Not completed — Did not return | 1 | 0
Not completed — Left before test | 0 | 1
Not completed — Left clinic early | 2 | 0
Period: 6-month Follow-up
Arm/Group | Rapid HIV Testing w/ Counseling (Group 1) | Rapid HIV Testing & Information Only (Group 2)
Started | 2505 | 2507
Completed | 2177 | 2179
Not Completed | 328 | 328
Not completed — Lost contact | 269 | 275
Not completed — Incarcerated | 37 | 32
Not completed — Withdrew consent | 14 | 15
Not completed — Death | 3 | 2
Not completed — Declined by Study Coordinator | 5 | 4

BASELINE CHARACTERISTICS:
Population: 6,239 patients approached provided consent to be screened. Of these, 5,028 were eligible (80.6%) and 5012 (99.5% of those eligible) were randomized; 16 screened eligible, but were not randomized due to: decision to decline (3), not returning (11), not testing with HIV/STD battery (1) and not completing baseline activities (1).
Groups:
- Total: Total of all reporting groups
Arm/Group | Rapid HIV Testing w/ Counseling (Group 1) | Rapid HIV Testing & Information Only (Group 2) | Total
Number analyzed (Participants) | 2505 | 2507 | 5012
Age, Customized [Number; unit: participants]
  <25 years | 1705 | 1727 | 3432
  >=25 years | 800 | 780 | 1580
Sex/Gender, Customized [Number; unit: participants]
  Male sex | 1655 | 1653 | 3308
  Female sex | 850 | 854 | 1704
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 1045 | 1053 | 2098
  Hispanic | 382 | 385 | 767
  White | 798 | 794 | 1592
  Other | 280 | 275 | 555
Region of Enrollment [Number; unit: participants]
  United States | 2505 | 2507 | 5012
Men who have sex with men (MSM), # [Number; unit: participants] — Men were classified as MSM if, at study intake, they reported any previous anal or oral sex with males or if on the baseline sexual risk behavior questions they reported having anal or oral sexwith another male at any time during the study. All men who did not meet the definition of MSM were classified as men who have sex with women.
  participants | 689 | 711 | 1400
Any STI, # [Number; unit: participants] | 1049 | 1092 | 2141
Any STI excluding trichomoniasis, # [Number; unit: participants] | 1016 | 1070 | 2086
Gonorrhea, # [Number; unit: participants] | 137 | 145 | 282
Chlamydia, # [Number; unit: participants] | 238 | 254 | 492
Trichomoniasis, # [Number; unit: participants] | 126 | 119 | 245
Syphilis, # [Number; unit: participants] | 28 | 35 | 63
HSV-2, # [Number; unit: participants] | 758 | 793 | 1551
HIV, # [Number; unit: participants] | 29 | 24 | 53
# of sex acts [Least Squares Mean (Standard Deviation); unit: sex acts] — Note that standard errors (not standard deviations) are presented below with the least squares means.
  sex acts | 34.6 (1.0809) | 33.4 (1.0431) | 34.0 (0.751)
# of unprotected sex acts [Least Squares Mean (Standard Deviation); unit: unprotected sex acts] — Note that standard errors (not standard deviations) are presented below with the least squares means.
  unprotected sex acts | 23.9 (0.9578) | 22.6 (0.9068) | 23.3 (0.6594)
# of partners [Least Squares Mean (Standard Deviation); unit: partners] — Note that standard errors (not standard deviations) are presented below with the least squares means.
  partners | 4.7 (0.1141) | 4.6 (0.1135) | 4.6 (0.08047)
# of unprotected partners [Least Squares Mean (Standard Deviation); unit: unprotected partners] — Note that standard errors (not standard deviations) are presented below with the least squares means.
  unprotected partners | 2.1 (0.05812) | 2.1 (0.05696) | 2.1 (0.04069)

OUTCOME MEASURES:

1. Primary Outcome: STI Incidence
Description: Composite STI incidence (Yes/No) at 6-month follow-up in which a person is considered positive for STIs if they are positive on any tested STI.
Time Frame: 6 months post randomization
Measure: Number; unit: participants
Arm/Group | Rapid HIV Testing w/ Counseling (Group 1) | Rapid HIV Testing & Information Only (Group 2)
Number analyzed (Participants) | 2039 | 2032
participants | 250 | 226
Statistical Analysis 1: Comparison: Rapid HIV Testing w/ Counseling (Group 1) vs Rapid HIV Testing & Information Only (Group 2); A total of 2039/2505 participants randomized to the counseling group and 2032/2507 to the information-only group had complete follow-up STI data. Cumulative STI incidence was 250/2039 (12.3%) in the counseling group and 226/2032 (11.1%) in the information-only group (aRR, 1.12; 95%CI, 0.94-1.33); Test type: Superiority or Other; Mantel Haenszel — In the statistical tests of all hypotheses and calculation of the presented risk ratios, we used multiple imputations of data sets with all 5012 cases. The aRRs reported are based on the multiply imputed data. Counts are based on the observed data; adjusted risk ratio (aRR) = 1.12, 95% CI 2-sided [0.94 to 1.33]

2. Secondary Outcome: Sexual Risk Behavior -- # of Sex Acts
Description: Self-reported continuous variables to determine number of (vaginal and/or anal) sex acts.
Time Frame: 6 months post randomization
Measure: Least Squares Mean (Standard Error); unit: sex acts
Arm/Group | Rapid HIV Testing w/ Counseling (Group 1) | Rapid HIV Testing & Information Only (Group 2)
Number analyzed (Participants) | 2505 | 2507
sex acts | 28.6 (1.1312) | 29.1 (1.1553)
Statistical Analysis 1: Comparison: Rapid HIV Testing w/ Counseling (Group 1) vs Rapid HIV Testing & Information Only (Group 2); Analyses of sexual risk behaviors used zero-inflated negative binomial regressions (ZINB) including treatment group, baseline level of the risk behavior, site, and randomization stratum. (ZINB regression was used instead of ANCOVA because the outcome variable had an excessive number of zeroes and over dispersion.) Adjusted incidence rate ratios (IRR) from the models are presented; Test type: Superiority or Other; Incidence rate ratio (IRR) = 0.99, 95% CI 2-sided [0.90 to 1.09] — In the statistical tests of all hypotheses and calculation of the presented IRR, we used multiple imputations of data sets with all 5012 cases. The adjusted IRRs reported are based on multiply imputed data. Counts are based on the observed data

3. Secondary Outcome: Sexual Risk Behavior -- # of Unprotected Sex Acts
Description: Self-reported continuous variables to determine number of unprotected (vaginal and/or anal) sex acts
Time Frame: 6 months post randomization
Measure: Least Squares Mean (Standard Error); unit: unprotected sex acts
Arm/Group | Rapid HIV Testing w/ Counseling (Group 1) | Rapid HIV Testing & Information Only (Group 2)
Number analyzed (Participants) | 2505 | 2507
unprotected sex acts | 17.4 (0.9791) | 18.3 (1.0381)
Statistical Analysis 1: Comparison: Rapid HIV Testing w/ Counseling (Group 1) vs Rapid HIV Testing & Information Only (Group 2); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Incidence Rate Ratio (IRR) = 0.98, 95% CI 2-sided [0.86 to 1.13] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Sexual Risk Behavior -- # of Partners
Description: Self-reported continuous variables to determine number of partners with whom the participant had (vaginal and/or anal) sex.
Time Frame: 6 months post randomization
Measure: Least Squares Mean (Standard Error); unit: partners
Arm/Group | Rapid HIV Testing w/ Counseling (Group 1) | Rapid HIV Testing & Information Only (Group 2)
Number analyzed (Participants) | 2505 | 2507
partners | 2.7 (0.07454) | 3.0 (0.08386)
Statistical Analysis 1: Comparison: Rapid HIV Testing w/ Counseling (Group 1) vs Rapid HIV Testing & Information Only (Group 2); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Incidence Rate Ratio (IRR) = 0.88, 95% CI 2-sided [0.82 to 0.94] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Sexual Risk Behavior -- # of Unprotected Partners
Description: Self-reported continuous variables to determine number of partners with whom the participant had unprotected (vaginal and/or anal) sex.
Time Frame: 6 months post randomization
Measure: Least Squares Mean (Standard Error); unit: unprotected partners
Arm/Group | Rapid HIV Testing w/ Counseling (Group 1) | Rapid HIV Testing & Information Only (Group 2)
Number analyzed (Participants) | 2505 | 2507
unprotected partners | 1.1 (0.03749) | 1.1 (0.03845)
Statistical Analysis 1: Comparison: Rapid HIV Testing w/ Counseling (Group 1) vs Rapid HIV Testing & Information Only (Group 2); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Incidence Rate Ratio (IRR) = 0.97, 95% CI 2-sided [0.90 to 1.05] — [estimate comment as in outcome 2, analysis 1]

6. Secondary Outcome: Sexual Risk Behavior -- # of Sex Acts With Substance Use
Description: Self-reported continuous variables to determine number of (vaginal and/or anal) sex acts in which the participant reported using substances before the sex act.
Time Frame: 6 months post randomization
Measure: Number; unit: sex acts with substance use
Arm/Group | Rapid HIV Testing w/ Counseling (Group 1) | Rapid HIV Testing & Information Only (Group 2)
Number analyzed (Participants) | 952 | 952
sex acts with substance use | 115 | 106
Statistical Analysis 1: Comparison: Rapid HIV Testing w/ Counseling (Group 1) vs Rapid HIV Testing & Information Only (Group 2); Test type: Superiority or Other; Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Adjusted Risk Ratio (aRR) = 1.14, 95% CI [0.89 to 1.46]

ADVERSE EVENTS:
Time Frame: Adverse events were captured post-randomization and were collected at each research visit. Other safety information is based on spontaneous reports and not specifically required by the study team.
Description: Only the following events were required for reporting as AEs: medical events that are directly related to the collection of the HIV and STI test samples (e.g. irritation at the testing site); additional AE were assessed based on report of untoward events that participant or investigator believes are a direct result of the study.
Arm/Group | Rapid HIV Testing w/ Counseling (Group 1) | Rapid HIV Testing & Information Only (Group 2)
Serious Adverse Events (participants affected / at risk) | 3/2505 | 2/2507
Other Adverse Events (participants affected / at risk) | 0/2505 | 0/2507
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rapid HIV Testing w/ Counseling (Group 1) (N=2505) | Rapid HIV Testing & Information Only (Group 2) (N=2507)
Death, cause unknown (General disorders) | 1 (1) | 0 (0) — "General disorders" selected as default; cause of death is unknown
victim of homicide, secondary to robbery (General disorders) | 1 (1) | 0 (0) — "General disorders" selected as default; cause is homicide
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Metastatic colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No